CLINICAL TRIAL: NCT00804856
Title: An Open Phase I/IIa Trial to Investigate the Maximum Tolerated Dose, Safety, Pharmacokinetics, and Efficacy of Intravenous BI 6727 as Monotherapy or in Combination With Subcutaneous Cytarabine in Patients With Acute Myeloid Leukaemia
Brief Title: Phase I/IIa Trial to Investigate BI 6727 (Volasertib) as Monotherapy or in Combination With Cytarabine in Acute Myeloid Leukaemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1230.4; 2008-003617-27 (EudraCT Number)
Record Dates: First submitted 2008-09-18; First posted 2008-12-09 (Estimated); Results first posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2022-12

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — BI 6727; Cytarabine

ARMS (15):
- Phase I Schedule A. Volasertib 150 mg+LDAC (Experimental): Volasertib 150 milligram (mg) administered by Intravenous Infusion (IV) over 60 minutes on Days 1 and 15 (28-day cycle) and Low-dose cytarabine (LDAC) 2x20mg per day administered by subcutaneous injection on days 1-10 of each 28 day treatment cycle.
  Interventions: Drug: Volasertib; Drug: Cytarabine
- Phase I Schedule A. Volasertib 200 mg+LDAC (Experimental): Volasertib 200 milligram (mg) administered by Intravenous Infusion (IV) over 60 minutes on Days 1 and 15 (28-day cycle) and Low-dose cytarabine (LDAC) 2x20mg per day administered by subcutaneous injection on days 1-10 of each 28 day treatment cycle.
  Interventions: Drug: Volasertib; Drug: Cytarabine
- Phase I Schedule A. Volasertib 250 mg+LDAC (Experimental): Volasertib 250 milligram (mg) administered by Intravenous Infusion (IV) over 60 minutes on Days 1 and 15 (28-day cycle) and Low-dose cytarabine (LDAC) 2x20mg per day administered by subcutaneous injection on days 1-10 of each 28 day treatment cycle.
  Interventions: Drug: Volasertib; Drug: Cytarabine
- Phase I Schedule A. Volasertib 300 mg+LDAC (Experimental): Volasertib 300 milligram (mg) administered by Intravenous Infusion (IV) over 60 minutes on Days 1 and 15 (28-day cycle) and Low-dose cytarabine (LDAC) 2x20mg per day administered by subcutaneous injection on days 1-10 of each 28 day treatment cycle.
  Interventions: Drug: Volasertib; Drug: Cytarabine
- Phase I Schedule A. Volasertib 350 mg+LDAC (Experimental): Volasertib 350 milligram (mg) administered by Intravenous Infusion (IV) over 60 minutes on Days 1 and 15 (28-day cycle) and Low-dose cytarabine (LDAC) 2x20mg per day administered by subcutaneous injection on days 1-10 of each 28 day treatment cycle.
  Interventions: Drug: Volasertib; Drug: Cytarabine
- Phase I Schedule A. Volasertib 400 mg+LDAC (Experimental): Volasertib 400 milligram (mg) administered by Intravenous Infusion (IV) over 60 minutes on Days 1 and 15 (28-day cycle) and Low-dose cytarabine (LDAC) 2x20mg per day administered by subcutaneous injection on days 1-10 of each 28 day treatment cycle.
  Interventions: Drug: Volasertib; Drug: Cytarabine
- Phase I Schedule B. Volasertib 150 mg (Experimental): Volasertib 150 milligram (mg) administered by Intravenous Infusion (IV) over 60 minutes on Days 1 and 15 (28-day cycle).
  Interventions: Drug: Volasertib
- Phase I Schedule B. Volasertib 200 mg (Experimental): Volasertib 200 milligram (mg) administered by Intravenous Infusion (IV) over 60 minutes on Days 1 and 15 (28-day cycle).
  Interventions: Drug: Volasertib
- Phase I Schedule B. Volasertib 350 mg (Experimental): Volasertib 350 milligram (mg) administered by Intravenous Infusion (IV) over 60 minutes on Days 1 and 15 (28-day cycle).
  Interventions: Drug: Volasertib
- Phase I Schedule B. Volasertib 400 mg (Experimental): Volasertib 400 milligram (mg) administered by Intravenous Infusion (IV) over 60 minutes on Days 1 and 15 (28-day cycle).
  Interventions: Drug: Volasertib
- Phase I Schedule B. Volasertib 450 mg (Experimental): Volasertib 450 milligram (mg) administered by Intravenous Infusion (IV) over 60 minutes on Days 1 and 15 (28-day cycle).
  Interventions: Drug: Volasertib
- Phase I Schedule B. Volasertib 500 mg (Experimental): Volasertib 500 milligram (mg) administered by Intravenous Infusion (IV) over 60 minutes on Days 1 and 15 (28-day cycle).
  Interventions: Drug: Volasertib
- Phase I Schedule B. Volasertib 550 mg (Experimental): Volasertib 550 milligram (mg) administered by Intravenous Infusion (IV) over 60 minutes on Days 1 and 15 (28-day cycle).
  Interventions: Drug: Volasertib
- Phase II Schedule C. LDAC (Active Comparator): Low-dose cytarabine (LDAC) monotherapy 2x20 milligram (mg) per day administered by subcutaneous injection on days 1-10 of each 28 days treatment cycle.
  Interventions: Drug: Cytarabine
- Phase II Schedule A. Volasertib 350 mg+LDAC (Experimental): Volasertib 350 milligram (mg) on Days 1 and 15 (28-day cycle) administered by Intravenous Infusion (IV) over 60 minutes and Low-dose cytarabine (LDAC) 2x20mg per day administered by subcutaneous injection on days 1-10 of each 28 days treatment cycle.
  Interventions: Drug: Volasertib; Drug: Cytarabine

INTERVENTIONS:
Drug: Volasertib — Volasertib administered by Intravenous Infusion (IV) over 60 minutes on Days 1 and 15 (28-day cycle).
  Arms: Phase I Schedule A. Volasertib 150 mg+LDAC; Phase I Schedule A. Volasertib 200 mg+LDAC; Phase I Schedule A. Volasertib 250 mg+LDAC; Phase I Schedule A. Volasertib 300 mg+LDAC; Phase I Schedule A. Volasertib 350 mg+LDAC; Phase I Schedule A. Volasertib 400 mg+LDAC; Phase I Schedule B. Volasertib 150 mg; Phase I Schedule B. Volasertib 200 mg; Phase I Schedule B. Volasertib 350 mg; Phase I Schedule B. Volasertib 400 mg; Phase I Schedule B. Volasertib 450 mg; Phase I Schedule B. Volasertib 500 mg; Phase I Schedule B. Volasertib 550 mg; Phase II Schedule A. Volasertib 350 mg+LDAC
Drug: Cytarabine — Low-dose cytarabine (LDAC) 2x20mg per day administered by subcutaneous injection on days 1-10 of each 28 day treatment cycle.
  Arms: Phase I Schedule A. Volasertib 150 mg+LDAC; Phase I Schedule A. Volasertib 200 mg+LDAC; Phase I Schedule A. Volasertib 250 mg+LDAC; Phase I Schedule A. Volasertib 300 mg+LDAC; Phase I Schedule A. Volasertib 350 mg+LDAC; Phase I Schedule A. Volasertib 400 mg+LDAC; Phase II Schedule A. Volasertib 350 mg+LDAC; Phase II Schedule C. LDAC

SUMMARY:
The trial will be performed in two parts, a phase I part and a phase IIa part. In the phase I part of the trial, BI 6727 will be investigated as monotherapy and in combination with low dose cytarabine (LD-Ara-C) in patients with relapsed/refractory AML that are not eligible for intensive treatment. The dose of BI 6727 will be escalated to determine the maximum tolerated dose (MTD) of BI 6727 monotherapy and BI 6727 in combination with LD-Ara-C in AML patients. In the phase IIa part, the combination of BI 6727 at MTD with LD-Ara-C and LD-Ara-C monotherapy will be investigated to explore the efficacy of the combination schedule in comparison to LD-Ara-C monotherapy in previously untreated AML patients that are not eligible for intensive treatment.

ELIGIBILITY:
Inclusion criteria:

Male or female adult with relapsed/refractory AML ineligible for intensive treatment (phase I part only) Male or female adult with previously untreated AML ineligible for intensive treatment (phase IIa part only) Confirmed diagnosis of AML according to the WHO definition (except for acute promyelocytic leukaemia, APL) Patient is eligible for LD-Ara-C treatment Life expectancy > 3 months Eastern co-operative oncology group (ECOG, R01-0787) performance score <=2 at screening Signed written informed consent consistent with international conference on harmonisation, good clinical practice (ICH-GCP) and local legislation

Exclusion criteria:

Previously untreated AML (phase I part only) Relapsed or treatment refractory AML (phase IIa part only) Patient with APL (AML subtype M3 according to the French-American-British (FAB) classification) Hypersensitivity to one of the trial drugs or the excipients Other malignancy requiring treatment Symptomatic central nervous system involvement Clinically relevant QT prolongation (e.g. long QT syndrome, QTcF>470 ms) Aspartate amino transferase (AST) or alanine amino transferase (ALT) greater than 2.5 times the upper limit of normal (ULN), or AST or ALT greater than 5 times the ULN in case of known leukaemia liver involvement Prothrombin time (PT) > 1.5 x ULN for subjects not on therapeutic vitamin K antagonists (phenprocoumon, warfarin) Bilirubin greater than 1.5 mg/dl (> 26 mcmol/L) Serum creatinine greater than 2.0 mg/dl Concomitant intercurrent illness, which would compromise the evaluation of efficacy or safety of the trial drug, e.g. active severe infection, unstable angina pectoris, cardiac arrhythmia or severe heart failure/cardiac insufficiency.

Psychiatric illness or social situation that would limit compliance with trial requirements Concomitant therapy, which is considered relevant for the evaluation of the efficacy or safety of the trial drug Contraindications for cytarabine treatment according to the SPC Female patients of childbearing potential who are sexually active and unwilling to use a medically acceptable method of contraception during the trial, i.e. combination of two forms of effective contraception (hormonal contraception, intrauterine device, condom with spermicide, etc.).

Male patients with partners of childbearing potential who are unwilling to use condoms in combination with a second medically acceptable method of contraception during the trial Pregnant or nursing female patients Patient unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2008-11-27 (Actual); Primary Completion 2012-03-09 (Actual); Study Completion 2021-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (27):
- LKH-Univ. Hospital Graz, Graz, Austria
- Belgium (3):
  - AZ Sint-Jan Brugge, Bruges
  - Brussels - UNIV Saint-Luc, Brussels
  - UZ Leuven, Leuven
- Canada (3):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Montreal General Hospital - McGill University Health Centre, Montreal, Quebec
  - CHUS Fleurimont, Sherbrooke, Quebec
- France (7):
  - HOP Clémenceau, Hémato, Caen, Caen
  - HOP, Centre Hospitalier René Dubos, Hémato, Paris, Cergy-Pontoise
  - HOP Dupuytren 1, Limoges
  - HOP Edouard Herriot, Lyon
  - CTR, fondation Paschetta, Hémato, Nice, Nice
  - HOP Saint-Louis, Paris
  - CTR Henri Becquerel, Rouen
- Germany (8):
  - Campus Virchow-Klinikum, Berlin, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Ulm, Ulm
- Italy (3):
  - A.O. Spedali Civili di Brescia, Brescia
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera Policlinico di Modena, Modena
- Norway (2):
  - Haukeland Universitetssykehus, Bergen
  - Oslo Universitetssykehus HF, Ullevål sykehus, Oslo

REFERENCES:
- [Derived] Dohner H, Lubbert M, Fiedler W, Fouillard L, Haaland A, Brandwein JM, Lepretre S, Reman O, Turlure P, Ottmann OG, Muller-Tidow C, Kramer A, Raffoux E, Dohner K, Schlenk RF, Voss F, Taube T, Fritsch H, Maertens J. Randomized, phase 2 trial of low-dose cytarabine with or without volasertib in AML patients not suitable for induction therapy. Blood. 2014 Aug 28;124(9):1426-33. doi: 10.1182/blood-2014-03-560557. Epub 2014 Jul 8. PMID 25006120
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open-label, randomized, dose escalation study. In this trial 180 patients were entered and randomised. However 3 patients were entered but not treated in Phase I and 2 patients were not treated in Phase II. Thus total 175 patients were treated in this trial.
Pre-assignment Details: Patients were assigned to two treatment schedules (A and B) in the phase I part of the trial (dose escalation phase to determine maximum tolerated dose (MTD)). In the phase IIa part of the trial (after MTD was determined), patients were randomised to two treatment schedules (A and C).
Period: Overall Study
Arm/Group | Phase I Schedule A. Volasertib 150 mg+LDAC | Phase I Schedule A. Volasertib 200 mg+LDAC | Phase I Schedule A. Volasertib 250 mg+LDAC | Phase I Schedule A. Volasertib 300 mg+LDAC | Phase I Schedule A. Volasertib 350 mg+LDAC | Phase I Schedule A. Volasertib 400 mg+LDAC | Phase I Schedule B. Volasertib 150 mg | Phase I Schedule B. Volasertib 200 mg | Phase I Schedule B. Volasertib 350 mg | Phase I Schedule B. Volasertib 400 mg | Phase I Schedule B. Volasertib 450 mg | Phase I Schedule B. Volasertib 500 mg | Phase I Schedule B. Volasertib 550 mg | Phase II Schedule C. LDAC | Phase II Schedule A. Volasertib 350 mg+LDAC
Started | 4 | 3 | 5 | 9 | 8 | 3 | 11 | 2 | 5 | 6 | 23 | 5 | 4 | 45 | 42
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 5 | 9 | 8 | 3 | 11 | 2 | 5 | 6 | 23 | 5 | 4 | 45 | 42
Not completed — Progressive Disease | 3 | 2 | 4 | 6 | 4 | 1 | 8 | 2 | 4 | 5 | 12 | 2 | 2 | 26 | 20
Not completed — Dose Limiting Toxicity (DLT) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other Adverse Event | 1 | 1 | 1 | 2 | 2 | 1 | 3 | 0 | 0 | 1 | 5 | 2 | 0 | 6 | 13
Not completed — Non compliance with protocol | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Refused to continue medication | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 5
Not completed — Other reason than listed above | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 10 | 3

BASELINE CHARACTERISTICS:
Population: Treated Set: All patients in Phase I who received at least a single dose of either Volasertib or LDAC, including patients who were replaced for any reason. For the Phase II part, the treated set (Phase II) was defined as all patients in Phase II who received at least a single dose of either Volasertib or LDAC.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Schedule A. Volasertib 150 mg+LDAC | Phase I Schedule A. Volasertib 200 mg+LDAC | Phase I Schedule A. Volasertib 250 mg+LDAC | Phase I Schedule A. Volasertib 300 mg+LDAC | Phase I Schedule A. Volasertib 350 mg+LDAC | Phase I Schedule A. Volasertib 400 mg+LDAC | Phase I Schedule B. Volasertib 150 mg | Phase I Schedule B. Volasertib 200 mg | Phase I Schedule B. Volasertib 350 mg | Phase I Schedule B. Volasertib 400 mg | Phase I Schedule B. Volasertib 450 mg | Phase I Schedule B. Volasertib 500 mg | Phase I Schedule B. Volasertib 550 mg | Phase II Schedule C. LDAC | Phase II Schedule A. Volasertib 350 mg+LDAC | Total
Number analyzed (Participants) | 4 | 3 | 5 | 9 | 8 | 3 | 11 | 2 | 5 | 6 | 23 | 5 | 4 | 45 | 42 | 175
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.5 (12.1) | 67.0 (3.0) | 71.2 (6.8) | 67.9 (12.0) | 72.5 (6.1) | 73.3 (7.6) | 73.5 (3.9) | 73.0 (4.2) | 70.6 (2.9) | 65.2 (20.1) | 68.2 (7.7) | 66.4 (7.3) | 69.8 (4.1) | 75.2 (5.5) | 75.6 (4.9) | 72.5 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2 | 3 | 3 | 1 | 3 | 1 | 3 | 2 | 16 | 1 | 3 | 20 | 19 | 79
  Male | 2 | 3 | 3 | 6 | 5 | 2 | 8 | 1 | 2 | 4 | 7 | 4 | 1 | 25 | 23 | 96
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 3 | 4 | 8 | 8 | 3 | 11 | 2 | 5 | 6 | 21 | 5 | 4 | 35 | 34 | 153
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 8 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of Volasertib in Combination With LDAC (Schedule A) and Volasertib Monotherapy (Schedule B)
Description: To determine the Maximum tolerated dose (MTD), dose escalation was conducted following the 3+3 design with de-escalation. The MTD was defined as the highest dose at which 6 patients had been treated and less than 2 patients experienced a Dose limiting toxicity (DLT) within the first cycle of treatment. The MTD was defined based on safety data from the first cycle only.
  DLT is defined as drug related Common terminology criteria for adverse events (CTCAE) grade ≥ 3 nonhaematological toxicity (excluding: untreated nausea, untreated vomiting, CTCAE grade 3 untreated diarrhoea, CTCAE grade 3 "febrile neutropenia" and CTCAE grade 3 "infection with grade 3 or 4 neutrophils").
  In patients with complete remission with incomplete blood count recovery (CRi) or partial remission (PR), persistent CTCAE grade 4 neutropenia or thrombocytopenia until three weeks after the end of the treatment cycle will be regarded a DLT.
Time Frame: First Treatment cycle, up to 28 days.
Population: Treated Set-phase I part: Treated Set was defined as all patients who received at least a single dose of either Volasertib (BI 6727) or LDAC (Low-Dose Cytarabine), including patients who were replaced for any reason.
Measure: Number; unit: milligram (mg)
Groups:
- Phase I Schedule A. Volasertib+LDAC: Patients were treated in the dose-escalation phase with Volasertib administered by Intravenous Infusion (IV) over 60 minutes on Days 1 and 15 (28-day cycle) and LDAC 2x20 milligram (mg) per day administered by subcutaneous injection on days 1-10 of each 28 day treatment cycle until the patient met criteria for stopping study medication during the MTD evaluation period.
- Phase I Schedule B. Volasertib: Patients were treated in the dose-escalation phase with Volasertib administered by Intravenous Infusion (IV) over 60 minutes on Days 1 and 15 (28-day cycle) until the patient met criteria for stopping study medication during the MTD evaluation period
Arm/Group | Phase I Schedule A. Volasertib+LDAC | Phase I Schedule B. Volasertib
Number analyzed (Participants) | 32 | 56
milligram (mg) | 350 | 450

2. Primary Outcome: Phase II: Number of Patients With Objective Response (Complete Remission (CR) + Complete Remission With Incomplete Blood Count Recovery (CRi))
Description: Phase II: Number of patients with Objective Response (Complete remission (CR) + Complete remission with incomplete blood count recovery (CRi)).
  Complete remission (CR): morphologically leukaemia-free state (i.e. bone marrow with <5% blasts by morphologic criteria and no Auer rods, no evidence of extramedullary leukaemia) and absolute neutrophil count ≥1,000/microliter (μL) and platelets >100,000/μL.
  Complete remission with incomplete blood count recovery ("incomplete" CR, CRi): all of the above criteria for CR were met except that neutrophils <1,000/μL or platelets <100,000/μL in the blood were not achieved.
Time Frame: The best overall response recorded during the time period from the start of the treatment until end of the treatment period, progression or death (whichever was earlier), up to 869 days.
Population: Treated set-phase II part: Treated Set was defined as all patients who received at least a single dose of either Volasertib or LDAC.
Measure: Count of Participants; unit: Participants
Groups:
- Phase II Schedule C. LDAC: Low-dose cytarabine (LDAC) monotherapy 2x20mg per day administered by subcutaneous injection on days 1-10 of each 28 days treatment cycle.
Arm/Group | Phase II Schedule C. LDAC | Phase II Schedule A. Volasertib 350 mg+LDAC
Number analyzed (Participants) | 45 | 42
Participants | 6 | 13
Statistical Analysis 1: Comparison: Phase II Schedule C. LDAC vs Phase II Schedule A. Volasertib 350 mg+LDAC; Analysis for Objective Response; Test type: Superiority or Other; p = 0.0523, Regression, Logistic; Odds Ratio (OR) = 2.91, 95% CI 2-sided [0.99 to 8.58] — Ratio calculated as Phase II Schedule A Volasertib 350mg+LDAC divided by Phase II Schedule C LDAC

3. Primary Outcome: Phase I: Number of Participants With Dose Limiting Toxicities (DLTs) in the First Cycle for the Determination of the Maximum Tolerated Dose (MTD)
Description: A DLT was defined as a drug related CTCAE (Common Toxicity Criteria for Adverse Events) Grade ≥3 non-haematological toxicity (excluding untreated nausea, untreated vomiting, Grade 3 untreated diarrhea, Grade 3 febrile neutropenia, and Grade 3 infection with Grade 3 or 4 neutrophils). In patients with CRi (Complete Remission with Incomplete Blood Count Recovery) or PR (Partial Remission), persistent Grade 4 neutropenia or thrombocytopenia for 3 weeks after the end of the treatment cycle was regarded as a DLT unless the respective Grade 4 cytopenia was preexistent. In patients who required platelet substitution to maintain a Grade <4 before treatment, a Grade 4 thrombocytopenia after treatment did not constitute a DLT.
Time Frame: First Treatment cycle, up to 28 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Total Phase I Combined. Schedule A.: Volasertib escalating dose on Days 1+15 (28-day cycle). Dose escalation in 50 mg steps up to 400 mg, with a starting dose of 400 mg. Volasertib administered by Intravenous Infusion (IV) over 60 minutes and LDAC 2x20mg per day administered by subcutaneous injection on days 1-10 of each 28 day treatment cycle.
- Total Phase I Combined. Schedule B.: Volasertib escalating dose on Days 1+15 (28-day cycle). Dose escalation in 50 mg steps from an initial starting dose of 150 mg. Dose was escalated up to 550 mg. Volasertib administered by Intravenous Infusion (IV) over 60 minutes.
Arm/Group | Phase I Schedule A. Volasertib 150 mg+LDAC | Phase I Schedule A. Volasertib 200 mg+LDAC | Phase I Schedule A. Volasertib 250 mg+LDAC | Phase I Schedule A. Volasertib 300 mg+LDAC | Phase I Schedule A. Volasertib 350 mg+LDAC | Phase I Schedule A. Volasertib 400 mg+LDAC | Total Phase I Combined. Schedule A. | Phase I Schedule B. Volasertib 150 mg | Phase I Schedule B. Volasertib 200 mg | Phase I Schedule B. Volasertib 350 mg | Phase I Schedule B. Volasertib 400 mg | Phase I Schedule B. Volasertib 450 mg | Phase I Schedule B. Volasertib 500 mg | Phase I Schedule B. Volasertib 550 mg | Total Phase I Combined. Schedule B.
Number analyzed (Participants) | 4 | 3 | 5 | 9 | 8 | 3 | 32 | 11 | 2 | 5 | 6 | 23 | 5 | 4 | 56
Participants | 0 | 0 | 0 | 1 | 1 | 2 | 4 | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 7

4. Secondary Outcome: Best Overall Response
Description: * CR
  * CR+CRi
  * Partial remission: CR except bone marrow (BM) contained ≥5% but <25% blasts (or ≤50% initial blasts), or <5% blasts in presence of Auer rods or abnormal morphology.
  * No change: survived ≥7 days (d) after 1st cycle with persistent leukemia in last peripheral blood smear or BM, or with persistent extramedullary disease, without further deterioration due to leukemia or increase of blasts in BM or peripheral blood.
  * Aplasia: survived ≥7d after 1st cycle, died whilst cytopenic, with last post-treatment BM result aplastic or hypoplastic and without leukemia blasts.
  * Indeterminate: survived <7 d after 1st cycle or survived ≥7d after 1st cycle, died with no persistent leukemia in peripheral smear but no post-treatment BM examination or did not complete 1st cycle.
  * Progressive disease: survived ≥7d after 1st cycle with increase of blast population in BM or peripheral blood or aggravation or new extramedullary disease or further deterioration or death due to leukemia.
Time Frame: as for outcome 2
Population: Treated Set-phase I part: Treated Set was defined as all patients who received at least a single dose of either Volasertib or LDAC, including patients who were replaced for any reason. Phase II part, the Treated Set was defined as all patients who received at least a single dose of either Volasertib or LDAC.
Measure: Count of Participants; unit: Participants
Groups:
- Total Phase I Combined. Schedule B.: Volasertib escalating dose on Days 1 and15 (28-day cycle). Dose escalation in 50 milligram (mg) steps from an initial starting dose of 150 mg; dose escalation stopped at 200 mg and then restarted from the MTD dose in Schedule A (350 mg); dose was escalated up to 550 mg. Volasertib administered by Intravenous Infusion (IV) over 60 minutes.
- Total Phase II Combined. Schedule A and C.: Volasertib escalating dose on Days 1 and 15 (28-day cycle). Dose escalation in 50 milligram (mg) steps up to 400 mg, with a starting dose of 150 mg. Volasertib 350 mg on Days 1+15 (28-day cycle) administered by Intravenous Infusion (IV) over 60 minutes and Low-dose cytarabine (LDAC) 2x20mg per day administered by subcutaneous injection on days 1-10 of each 28 day treatment cycle.
Arm/Group | Phase I Schedule A. Volasertib 150 mg+LDAC | Phase I Schedule A. Volasertib 200 mg+LDAC | Phase I Schedule A. Volasertib 250 mg+LDAC | Phase I Schedule A. Volasertib 300 mg+LDAC | Phase I Schedule A. Volasertib 350 mg+LDAC | Phase I Schedule A. Volasertib 400 mg+LDAC | Total Phase I Combined. Schedule A. | Phase I Schedule B. Volasertib 150 mg | Phase I Schedule B. Volasertib 200 mg | Phase I Schedule B. Volasertib 350 mg | Phase I Schedule B. Volasertib 400 mg | Phase I Schedule B. Volasertib 450 mg | Phase I Schedule B. Volasertib 500 mg | Phase I Schedule B. Volasertib 550 mg | Total Phase I Combined. Schedule B. | Phase II Schedule C. LDAC | Phase II Schedule A. Volasertib 350 mg+LDAC | Total Phase II Combined. Schedule A and C.
Number analyzed (Participants) | 4 | 3 | 5 | 9 | 8 | 3 | 32 | 11 | 2 | 5 | 6 | 23 | 5 | 4 | 56 | 45 | 42 | 87
Participants
  Complete remission | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 9
  CRi | 0 | 2 | 0 | 1 | 1 | 0 | 4 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 5 | 3 | 7 | 10
  Partial remission | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 4 | 2 | 2 | 4
  No change | 2 | 1 | 2 | 1 | 1 | 1 | 8 | 4 | 0 | 2 | 2 | 7 | 3 | 0 | 18 | 18 | 15 | 33
  Aplasia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 6 | 0 | 0 | 0
  Indeterminate | 0 | 0 | 0 | 2 | 3 | 1 | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 5 | 8
  Progressive disease | 2 | 0 | 1 | 3 | 3 | 1 | 10 | 6 | 2 | 1 | 1 | 7 | 1 | 1 | 19 | 14 | 7 | 21
  Not evaluable | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3 | 2 | 0 | 2
  Missing | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Phase I: Number of Patients With Objective Response: Complete Remission or Complete Remission With Incomplete Blood Count Recovery (CR+CRi)
Description: Phase I: Number of patients with Objective Response (Complete remission (CR) + Complete remission with incomplete blood count recovery (CRi)).
  Complete remission (CR): morphologically leukaemia-free state (i.e. bone marrow with <5% blasts by morphologic criteria and no Auer rods, no evidence of extramedullary leukaemia) and absolute neutrophil count ≥1,000/microliter (μL) and platelets >100,000/μL.
  Complete remission with incomplete blood count recovery ("incomplete" CR, CRi): all of the above criteria for CR were met except that neutrophils <1,000/μL or platelets <100,000/μL in the blood were not achieved.
Time Frame: The best overall response recorded during the time period from the start of the treatment until end of the treatment period, progression or death (whichever was earlier), up to 594 days.
Population: Treated Set-phase I part: Treated Set was defined as all patients who received at least a single dose of either Volasertib or LDAC, including patients who were replaced for any reason.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Schedule A. Volasertib 150 mg+LDAC | Phase I Schedule A. Volasertib 200 mg+LDAC | Phase I Schedule A. Volasertib 250 mg+LDAC | Phase I Schedule A. Volasertib 300 mg+LDAC | Phase I Schedule A. Volasertib 350 mg+LDAC | Phase I Schedule A. Volasertib 400 mg+LDAC | Total Phase I Combined. Schedule A. | Phase I Schedule B. Volasertib 150 mg | Phase I Schedule B. Volasertib 200 mg | Phase I Schedule B. Volasertib 350 mg | Phase I Schedule B. Volasertib 400 mg | Phase I Schedule B. Volasertib 450 mg | Phase I Schedule B. Volasertib 500 mg | Phase I Schedule B. Volasertib 550 mg | Total Phase I Combined. Schedule B.
Number analyzed (Participants) | 4 | 3 | 5 | 9 | 8 | 3 | 32 | 11 | 2 | 5 | 6 | 23 | 5 | 4 | 56
Participants | 0 | 2 | 2 | 1 | 1 | 0 | 6 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 5

6. Secondary Outcome: Phase II: Event Free Survival
Description: Event-free survival (EFS) [days] was the shortest duration of the following: (a) Date of assessment indicating PD on the response page of the eCRF (Electronic Case Report Form) - date of randomisation + 1 day (b) Date of assessment indicating clinical progressive disease (PD) on the disease or responses pages of the of eCRF- date of randomisation + 1 day (c) Date of assessment indicating PD on the patient status page of the eCRF - date of randomisation +1 day (for patients who had not been censored before this time point) (d) Death date - date of randomisation +1 day Patients not being assessed PD, clinical PD, or death during the trial were censored.
  EFS was analysed with the Kaplan-Meier method for each of the treatment arms.
Time Frame: The patients that entered the trial, and measured from the date of randomization to the date of disease progression (treatment failure), relapse or death from any cause, whichever occurred first, up to 1000 days..
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Phase II Schedule C. LDAC | Phase II Schedule A. Volasertib 350 mg+LDAC
Number analyzed (Participants) | 45 | 42
Days | 69.0 [27 to 215] | 169.0 [39 to 470]
Statistical Analysis 1: Comparison: Phase II Schedule C. LDAC vs Phase II Schedule A. Volasertib 350 mg+LDAC; An exploratory (non-stratified) logrank test was used to compare the different treatment arms; Test type: Superiority or Other; p = 0.0208, Log Rank; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.35 to 0.92] — Ratio calculated as Phase II Schedule A Volasertib 350mg+LDAC divided by Phase II Schedule C LDAC

7. Secondary Outcome: Phase II: Overall Survival
Description: Overall survival [days] = (date of death - date of randomisation + 1 day), for patients with known date of death. Overall survival (censored) [days] = (date of last trial visit or follow-up - date of randomisation + 1 day), for patients who were still alive at time of database lock.
  Overall survival (OS) was analysed with the Kaplan-Meier method for each of the treatment arms.
Time Frame: The patients that entered the trial, and measured from the date of randomisation until death from any cause, up to 1100 days..
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Phase II Schedule C. LDAC | Phase II Schedule A. Volasertib 350 mg+LDAC
Number analyzed (Participants) | 45 | 42
Days | 158.0 [78 to 347] | 245.0 [73 to 689]
Statistical Analysis 1: Comparison: Phase II Schedule C. LDAC vs Phase II Schedule A. Volasertib 350 mg+LDAC; An exploratory (non-stratified) logrank test was used to compare the different treatment arms; Test type: Superiority or Other; p = 0.0465, Log Rank; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.40 to 1.00] — Ratio calculated as Phase II Schedule A Volasertib 350mg+LDAC divided by Phase II Schedule C LDAC

8. Secondary Outcome: Phase II: Relapse - Free Survival
Description: Relapse-free survival [days] = (date of first recurrence of disease or death after entering the trial - date of first occurrence of CR or CRi after entering the trial+ 1 day) for patients with a recurrence (this value should be positive).
  Relapse-free survival (censored) [days] = (date of last trial visit or follow-up - date of first occurrence of CR or CRi after entering the trial + 1 day) for patients who did not experience recurrence of disease or death at the time of analysis.
Time Frame: The patients who achieved CR or CRi, and was measured from the date of attaining CR or CRi until the date of disease recurrence or death from any cause, whichever occurred first, up to 900 days.
Population: Patients in Treated Set-Phase II with objective response. Treated Set-Phase II part: Treated Set was defined as all patients who received at least a single dose of either Volasertib or LDAC.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Phase II Schedule C. LDAC | Phase II Schedule A. Volasertib 350 mg+LDAC
Number analyzed (Participants) | 6 | 13
Days | 304.0 [113 to 367] | 563.0 [427 to NA] — 25% quartile not reached, not enough events occurred.

9. Secondary Outcome: Phase II: Remission Duration
Description: Remission duration analysis was defined only for patients who achieved Complete remission (CR) or Complete remission with incomplete blood count recovery (CRi), and was measured from the date of attaining CR or CRi until the date of disease recurrence (relapse). For patients who died without report of relapse, remission duration was censored on the date of death, regardless of cause.
Time Frame: The patients who achieved CR or CRi, and was measured from the date of attaining CR or CRi until the date of disease recurrence (relapse), up to 900 days.
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Phase II Schedule C. LDAC | Phase II Schedule A. Volasertib 350 mg+LDAC
Number analyzed (Participants) | 6 | 13
Days | 367.0 [113 to 367] | 687.0 [427 to NA] — 25% quartile not reached, not enough events occurred.

10. Secondary Outcome: Phase II: Time to Remission
Description: Time to remission [days] = (date of first occurrence of CR or CRi after entering the trial-date of randomisation + 1 day) for patients with an objective response.
Time Frame: The patients who achieved CR or CRi, and was measured from the date of attaining CR or CRi until the date of disease recurrence (relapse), up to 158 days.
Population: as for outcome 8
Measure: Median (Full Range); unit: Days
Arm/Group | Phase II Schedule C. LDAC | Phase II Schedule A. Volasertib 350 mg+LDAC
Number analyzed (Participants) | 6 | 13
Days | 63.5 [30 to 125] | 71.0 [29 to 158]

11. Secondary Outcome: Best Eastern Co-operative Oncology Group (ECOG) Performance Score From Baseline Until End of Treatment
Description: ECOG performance score change from baseline to last visit of last cycle = ECOG performance score at last visit of the last cycle - ECOG performance score at baseline. ECOG performance score changes from baseline were also categorised on a 3-point categorical scale: deteriorated (-1), unchanged (0), and improved (1). The number of participants for category of ECOG score change is reported.
Time Frame: Baseline and End of Treatment (up to 869 days).
Population: Treated Set-Phase I part: Treated Set was defined as all patients who received at least a single dose of either Volasertib or LDAC, including patients who were replaced for any reason. Phase II part, the Treated Set was defined as all patients who received at least a single dose of either Volasertib or LDAC. Only participants with non-missing values are reported.
Measure: Count of Participants; unit: Participants
Groups:
- Total Phase I Combined. Schedule A.: Volasertib escalating dose on Days 1 and 15 (28-day cycle). Dose escalation in 50 milligram (mg) steps up to 400 mg, with a starting dose of 400 mg. Volasertib administered by Intravenous Infusion (IV) over 60 minutes and Low-dose cytarabine (LDAC) 2x20mg per day administered by subcutaneous injection on days 1-10 of each 28 day treatment cycle.
- Total Phase I Comined. Schedule B.: Volasertib escalating dose on Days 1 and 15 (28-day cycle). Dose escalation in 50 milligram (mg) steps from an initial starting dose of 550 mg. Dose was escalated up to 550 mg. Volasertib administered by Intravenous Infusion (IV) over 60 minutes.
- Total Phase II. Schedule A and C.: Volasertib escalating dose on Days 1 and 15 (28-day cycle). Dose escalation in 50 milligram (mg) steps up to 400 mg, with a starting dose of 150 mg. Volasertib 350 mg on Days 1+15 (28-day cycle) administered by Intravenous Infusion (IV) over 60 minutes and Low-dose cytarabine (LDAC) 2x20mg per day administered by subcutaneous injection on days 1-10 of each 28 day treatment cycle.
Arm/Group | Phase I Schedule A. Volasertib 150 mg+LDAC | Phase I Schedule A. Volasertib 200 mg+LDAC | Phase I Schedule A. Volasertib 250 mg+LDAC | Phase I Schedule A. Volasertib 300 mg+LDAC | Phase I Schedule A. Volasertib 350 mg+LDAC | Phase I Schedule A. Volasertib 400 mg+LDAC | Total Phase I Combined. Schedule A. | Phase I Schedule B. Volasertib 150 mg | Phase I Schedule B. Volasertib 200 mg | Phase I Schedule B. Volasertib 350 mg | Phase I Schedule B. Volasertib 400 mg | Phase I Schedule B. Volasertib 450 mg | Phase I Schedule B. Volasertib 500 mg | Phase I Schedule B. Volasertib 550 mg | Total Phase I Comined. Schedule B. | Phase II Schedule C. LDAC | Phase II Schedule A. Volasertib 350 mg+LDAC | Total Phase II. Schedule A and C.
Number analyzed (Participants) | 4 | 3 | 5 | 5 | 8 | 2 | 27 | 10 | 2 | 5 | 6 | 22 | 5 | 3 | 53 | 42 | 39 | 81
Participants
  Unchanged | 3 | 1 | 5 | 2 | 5 | 1 | 17 | 9 | 1 | 0 | 4 | 14 | 2 | 3 | 33 | 22 | 15 | 37
  Improved | 0 | 2 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 6 | 8 | 13 | 21
  Deteriorated | 1 | 0 | 0 | 2 | 3 | 1 | 7 | 1 | 1 | 4 | 1 | 5 | 2 | 0 | 14 | 12 | 11 | 23

12. Secondary Outcome: Total Clearance (CL) of Volasertib in Plasma After i.v (Intravenous) Administration of Volasertib
Description: Total Clearance (CL) of Volasertib in Plasma after Intravenous (i.v.) Administration of Volasertib.
Time Frame: Cycle 1: -0:05 hour (h), 0:30h, 1:00h, 1:30h, 2h, 3h, 4h, 24h, 96h, 216h, 335:55h, 336:30h, 337h, 337:30h, 338h, 339h, 340h, 648h after first drug administration.
Population: Pharmacokinetic (PK) set which included all patients in the treated set who had at least 1 evaluable blood sample during cycle 1. Phase I Schedule B Volasertib 200mg+LDAC was not analysed as there was not enough plasma concentrations at the terminal phase of the curve to calculate the half-life for one of the two subjects.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: millilitre/minute (mL/min)
Groups:
- Phase II Schedule A. Volasertib 350 mg+LDAC.: Volasertib 350 mg on Days 1+15 (28-day cycle) administered by Intravenous Infusion (IV) over 60 minutes and LDAC 2x20mg per day administered by subcutaneous injection on days 1-10 of each 28 day treatment cycle.
Arm/Group | Phase I Schedule A. Volasertib 150 mg+LDAC | Phase I Schedule A. Volasertib 200 mg+LDAC | Phase I Schedule A. Volasertib 250 mg+LDAC | Phase I Schedule A. Volasertib 300 mg+LDAC | Phase I Schedule A. Volasertib 350 mg+LDAC | Phase I Schedule A. Volasertib 400 mg+LDAC | Phase I Schedule B. Volasertib 150 mg | Phase I Schedule B. Volasertib 200 mg | Phase I Schedule B. Volasertib 350 mg | Phase I Schedule B. Volasertib 400 mg | Phase I Schedule B. Volasertib 450 mg | Phase I Schedule B. Volasertib 500 mg | Phase I Schedule B. Volasertib 550 mg | Phase II Schedule A. Volasertib 350 mg+LDAC.
Number analyzed (Participants) | 4 | 3 | 5 | 8 | 8 | 3 | 10 | 1 | 5 | 6 | 22 | 5 | 3 | 31
millilitre/minute (mL/min) | 1280 (52.8) | 972 (26.6) | 864 (27.6) | 1150 (34.4) | 1000 (36.2) | 852 (49.6) | 1330 (29.3) | NA (NA) — Not calculable with one subject | 810 (35.1) | 1120 (62.1) | 920 (36.2) | 1140 (38.5) | 939 (93.2) | 897 (42.8)

13. Secondary Outcome: Apparent Volume of Distribution of Volasertib at Steady State (VSS)
Description: Apparent Volume of Distribution of volasertib at steady state (VSS) following Intravenous (i.v.) administration.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Phase I Schedule A. Volasertib 150 mg+LDAC | Phase I Schedule A. Volasertib 200 mg+LDAC | Phase I Schedule A. Volasertib 250 mg+LDAC | Phase I Schedule A. Volasertib 300 mg+LDAC | Phase I Schedule A. Volasertib 350 mg+LDAC | Phase I Schedule A. Volasertib 400 mg+LDAC | Phase I Schedule B. Volasertib 150 mg | Phase I Schedule B. Volasertib 200 mg | Phase I Schedule B. Volasertib 350 mg | Phase I Schedule B. Volasertib 400 mg | Phase I Schedule B. Volasertib 450 mg | Phase I Schedule B. Volasertib 500 mg | Phase I Schedule B. Volasertib 550 mg | Phase II Schedule A. Volasertib 350 mg+LDAC.
Number analyzed (Participants) | 4 | 3 | 5 | 8 | 8 | 3 | 10 | 1 | 5 | 6 | 22 | 5 | 3 | 31
Liter (L) | 10600 (111.0) | 8640 (14.1) | 7000 (26.6) | 6320 (35.9) | 5270 (58.2) | 4830 (56.7) | 10300 (36.3) | NA (NA) — Not calculable with one subject | 5800 (35.1) | 7150 (70.6) | 5740 (38.7) | 6360 (50.1) | 5680 (81.9) | 6130 (42.0)

14. Secondary Outcome: Dose Normalized Maximum Measured Concentration of Cytarabine in Plasma (Cmax, Norm)
Description: Cmax, norm: Maximum measured concentration of Cytarabine in plasma. The dose normalisation was done by dividing by the dose applied. Unit: nanogram/milliliter/milligram: ((ng/mL)/mg). Dose groups of Phase I were combined by dose normalizing as pre specified in the study protocol.
Time Frame: as for outcome 12
Population: Pharmacokinetic (PK) set which included all patients in the treated set who had at least 1 evaluable blood sample during cycle 1, Only participants with non-missing values are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng/mL)/mg
Groups:
- Dose Normalized Volasertib+LDAC(Phase I,Schedule A). 150 to 400 mg Volasertib.: Volasertib 150 to 400 milligram (mg) administered by Intravenous Infusion (IV) over 60 minutes on Days 1 and 15 (28-day cycle) and Low-dose cytarabine (LDAC) 2x20mg per day administered by subcutaneous injection on days 1-10 of each 28 day treatment cycle. Dose groups of Phase I were combined by dose normalizing as pre specified in the study protocol.
- Dose Normalized Volasertib+LDAC (Schedule A). Phase II. 350 mg Volasertib.: Volasertib 350 milligram (mg) on Days 1 and 15 (28-day cycle) administered by Intravenous Infusion (IV) over 60 minutes and Low-dose cytarabine (LDAC) 2x20mg per day administered by subcutaneous injection on days 1-10 of each 28 days treatment cycle.
- Dose Normalized LDAC (Schedule C). Phase II. LDAC Monotherapy.: Low-dose cytarabine (LDAC) monotherapy 2x20 milligram (mg) per day administered by subcutaneous injection on days 1-10 of each 28 days treatment cycle.
Arm/Group | Dose Normalized Volasertib+LDAC(Phase I,Schedule A). 150 to 400 mg Volasertib. | Dose Normalized Volasertib+LDAC (Schedule A). Phase II. 350 mg Volasertib. | Dose Normalized LDAC (Schedule C). Phase II. LDAC Monotherapy.
Number analyzed (Participants) | 32 | 41 | 40
(ng/mL)/mg | 2.92 (61.3) | 2.83 (52.8) | 2.36 (77.6)

15. Secondary Outcome: Dose Normalized Area Under the Concentration-Time Curve of Cytarabine in Plasma Over the Time Interval From 0 Extrapolated up to 4 Hours
Description: AUC0-4,norm: Area under the concentration-time curve of Cytarabine in plasma over the time interval from zero extrapolated to 4 hours. The dose normalisation was done by dividing by dose applied. Unit: nanogram*hour/milliliter/milligram: ((ng*h/mL)/mg).
  Dose groups of Phase I were combined by dose normalizing as pre specified in the study protocol.
Time Frame: Cycle 1: -0:05 hour (h), 0:30h, 1:00h, 1:30h, 2h, 3h, 4h after first drug administration.
Population: Pharmacokinetic (PK) set which included all patients in the treated set who had at least 1 evaluable blood sample during cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng*h/mL)/mg
Groups:
- Dose Normalized LDAC (Schedule C). Phase II. LDAC Monotherapy.: Low-dose cytarabine (LDAC) monotherapy 2x20 milligram (mg) per day administered by subcutaneous injection on days 1-10 of each 28 days treatment.
Arm/Group | Dose Normalized Volasertib+LDAC(Phase I,Schedule A). 150 to 400 mg Volasertib. | Dose Normalized Volasertib+LDAC (Schedule A). Phase II. 350 mg Volasertib. | Dose Normalized LDAC (Schedule C). Phase II. LDAC Monotherapy.
Number analyzed (Participants) | 32 | 41 | 40
(ng*h/mL)/mg | 3.84 (30.6) | 4.00 (35.6) | 3.94 (43.8)

16. Secondary Outcome: Absolute QTcF (QT Interval Corrected for Heart Rate Using Fridericia's Formula) Intervals
Description: ECG (Electro Cardio Gram) Measurements: Absolute QTcF (QT Interval (interval from the beginning of the QRS complex to the end of the T wave) Corrected for Heart Rate Using Fridericia's Formula) Intervals. The 350 mg + LDAC arm of phase I and II were combined into one arm to provide maximum information on QT changes and presented together with the Phase I schedule B 450 mg arm, as pre specified in the study protocol.
Time Frame: Baseline (Days -14 to -1) and day 1 (1 hour and 24 hours) after start of infusion.
Population: Treated Set-Phase I part: Treated Set was defined as all patients who received at least a single dose of either Volasertib or LDAC, including patients who were replaced for any reason. Only participants with non-missing values are reported.
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Groups:
- Phase I+II Volasertib 350 mg+LDAC: Phase I+II: Volasertib 350 milligram (mg) administered by Intravenous Infusion (IV) over 60 minutes on Days 1 and 15 (28-day cycle) and Low-dose cytarabine (LDAC) 2x20mg per day administered by subcutaneous injection on days 1-10 of each 28 day treatment cycle.
Arm/Group | Phase I+II Volasertib 350 mg+LDAC | Phase I Schedule B. Volasertib 450 mg
Number analyzed (Participants) | 50 | 23
milliseconds (ms)
  Individual baseline | 411.6 (20.7) | 412.4 (18.7)
  1 hour after start of infusion: number analyzed (Participants) | 49 | 22
  1 hour after start of infusion | 430.0 (20.4) | 441.1 (20.0)
  24 hour after start of infusion: number analyzed (Participants) | 49 | 23
  24 hour after start of infusion | 414.0 (21.3) | 411.9 (18.4)

17. Secondary Outcome: QTcF (QT Interval Corrected for Heart Rate Using Fridericia's Formula) Change From Baseline at Cycle 1
Description: ECG Measurements: QTcF (QT Interval (interval from the beginning of the QRS complex to the end of the T wave) changes from baseline at each time point: The QTcF post baseline measurement obtained at time t minus baseline QTcF measurement. The 350 mg + LDAC arm of phase I and II were combined into one arm to provide maximum information on QT changes and presented together with the Phase I schedule B 450 mg arm, as pre specified in the study protocol.
Time Frame: Baseline (Days -14 to -1) and day 1 (1 hour and 24 hours) after start of infusion.
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: millisecond (ms)
Groups:
- Phase I+II, Volasertib 350 mg+LDAC: Phase I+II: Volasertib 350 mg administered by Intravenous Infusion (IV) over 60 minutes on Days 1+15 (28-day cycle) and LDAC 2x20mg per day administered by subcutaneous injection on days 1-10 of each 28 day treatment cycle.
Arm/Group | Phase I+II, Volasertib 350 mg+LDAC | Phase I Schedule B. Volasertib 450 mg
Number analyzed (Participants) | 50 | 23
millisecond (ms)
  Change from baseline after 1 hour: number analyzed (Participants) | 49 | 22
  Change from baseline after 1 hour | 18.5 (10.4) | 29.6 (8.1)
  Change from baseline after 24 hour: number analyzed (Participants) | 49 | 23
  Change from baseline after 24 hour | 1.9 (10.5) | -0.5 (9.8)

18. Secondary Outcome: Phase I Schedule A: Number of Participants With Adverse Events (AEs) Graded According to Common Terminology Criteria for Adverse Events (CTCAE), Based on the Number of Patients With AEs With CTCAE Grade ≥3 During Cycle 1
Description: Number of patients with AEs following in the categories 3 (severe AE), 4 (life-threatening or disabling AE), 5 (death related AE) of CTCAE is reported.
Time Frame: First treatment cycle, up to 28 days.
Population: Treated set-Phase I part: Treated set was defined as all patients in Phase I who received at least a single dose of either Volasertib or LDAC, including patients who were replaced for any reason.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Schedule A. Volasertib 150 mg+LDAC | Phase I Schedule A. Volasertib 200 mg+LDAC | Phase I Schedule A. Volasertib 250 mg+LDAC | Phase I Schedule A. Volasertib 300 mg+LDAC | Phase I Schedule A. Volasertib 350 mg+LDAC | Phase I Schedule A. Volasertib 400 mg+LDAC | Total Phase I Combined. Schedule A.
Number analyzed (Participants) | 4 | 3 | 5 | 9 | 8 | 3 | 32
Participants
  Grade 3 | 0 | 0 | 1 | 1 | 2 | 1 | 5
  Grade 4 | 2 | 3 | 3 | 5 | 3 | 1 | 17
  Grade 5 | 0 | 0 | 0 | 3 | 2 | 1 | 6

19. Secondary Outcome: Phase I Schedule B: Number of Participants With Adverse Events (AEs) Graded According to Common Terminology Criteria for Adverse Events (CTCAE), Based on the Number of Patients With AEs With CTCAE Grade ≥3 During Cycle 1
Description: as for outcome 18
Time Frame: First treatment cycle, up to 28 days.
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Groups:
- Total Phase I Schedule B.: Volasertib escalating dose on Days 1+15 (28-day cycle). Dose escalation in 50 mg steps from an initial starting dose of 150 mg. Dose was escalated up to 550 mg. Volasertib administered by Intravenous Infusion (IV) over 60 minutes.
Arm/Group | Phase I Schedule B. Volasertib 150 mg | Phase I Schedule B. Volasertib 200 mg | Phase I Schedule B. Volasertib 350 mg | Phase I Schedule B. Volasertib 400 mg | Phase I Schedule B. Volasertib 450 mg | Phase I Schedule B. Volasertib 500 mg | Phase I Schedule B. Volasertib 550 mg | Total Phase I Schedule B.
Number analyzed (Participants) | 11 | 2 | 5 | 6 | 23 | 5 | 4 | 56
Participants
  Grade 3 | 5 | 0 | 1 | 0 | 5 | 0 | 0 | 11
  Grade 4 | 4 | 1 | 3 | 4 | 14 | 1 | 3 | 30
  Grade 5 | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 6

20. Secondary Outcome: Phase I Schedule A: Number of Participants With Adverse Events (AEs) Graded According to Common Terminology Criteria for Adverse Events (CTCAE), Based on the Number of Patients With AEs With CTCAE Grade ≥3 During All Cycles
Description: as for outcome 18
Time Frame: From first drug administration until 21 days after the last trial drug administration in the last treatment cycle, up to 615 days.
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Schedule A. Volasertib 150 mg+LDAC | Phase I Schedule A. Volasertib 200 mg+LDAC | Phase I Schedule A. Volasertib 250 mg+LDAC | Phase I Schedule A. Volasertib 300 mg+LDAC | Phase I Schedule A. Volasertib 350 mg+LDAC | Phase I Schedule A. Volasertib 400 mg+LDAC | Total Phase I Combined. Schedule A.
Number analyzed (Participants) | 4 | 3 | 5 | 9 | 8 | 3 | 32
Participants
  Grade 3 | 1 | 0 | 0 | 1 | 2 | 1 | 5
  Grade 4 | 1 | 3 | 5 | 5 | 3 | 1 | 18
  Grade 5 | 1 | 0 | 0 | 3 | 2 | 1 | 7

21. Secondary Outcome: Phase I Schedule B: Number of Participants With Adverse Events (AEs) Graded According to Common Terminology Criteria for Adverse Events (CTCAE), Based on the Number of Patients With AEs With CTCAE Grade ≥3 During All Cycles
Description: as for outcome 18
Time Frame: From first drug administration until 21 days after the last trial drug administration in the last treatment cycle, up to 597 days.
Population: Treated set-Phase I part: the treated set was defined as all patients in Phase I who received at least a single dose of either Volasertib or LDAC, including patients who were replaced for any reason.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Schedule B. Volasertib 150 mg | Phase I Schedule B. Volasertib 200 mg | Phase I Schedule B. Volasertib 350 mg | Phase I Schedule B. Volasertib 400 mg | Phase I Schedule B. Volasertib 450 mg | Phase I Schedule B. Volasertib 500 mg | Phase I Schedule B. Volasertib 550 mg | Total Phase I Schedule B.
Number analyzed (Participants) | 11 | 2 | 5 | 6 | 23 | 5 | 4 | 56
Participants
  Grade 3 | 5 | 0 | 1 | 0 | 3 | 0 | 0 | 9
  Grade 4 | 4 | 1 | 3 | 5 | 15 | 1 | 3 | 32
  Grade 5 | 2 | 1 | 0 | 0 | 3 | 2 | 1 | 9

22. Secondary Outcome: Phase II: Number of Participants With Adverse Events (AEs) Graded According to Common Terminology Criteria for Adverse Events (CTCAE), Based on the Number of Patients With AEs With CTCAE Grade ≥3 During All Cycles
Description: Number of patients with AEs following in the in the categories 3 (severe AE), 4 (life-threatening or disabling AE), 5 (death related AE) of CTCAE is reported.
Time Frame: From first drug administration until 21 days after the last trial drug administration in the last treatment cycle, up to 890 days.
Population: Treated set-Phase II part: the treated set (Phase II) was defined as all patients in Phase II who received at least a single dose of either Volasertib or LDAC.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II Schedule C. LDAC | Phase II Schedule A. Volasertib 350 mg+LDAC
Number analyzed (Participants) | 45 | 42
Participants
  Grade 3 | 13 | 12
  Grade 4 | 13 | 20
  Grade 5 | 6 | 8

ADVERSE EVENTS:
Time Frame: From first drug administration until 21 days after the last trial drug administration in the last treatment cycle, up to 3325 days.
Description: Treated Set-phase I part: Treated Set was defined as all patients who received at least a single dose of either Volasertib or Low-dose cytarabine (LDAC), including patients who were replaced for any reason. Phase II part, the Treated Set was defined as all patients who received at least a single dose of either Volasertib or LDAC.
Groups:
- Phase II Schedule A. Volasertib 350 mg+LDAC: Volasertib 350 milligram (mg) administered by Intravenous Infusion (IV) over 60 minutes on Days 1 and 15 (28-day cycle) and Low-dose cytarabine (LDAC) 2x20mg per day administered by subcutaneous injection on days 1-10 of each 28 day treatment cycle.
- Phase I Schedule B. Volasertib 400 mg: Phase I Schedule B. Volasertib 400 mg Volasertib 400 milligram (mg) administered by Intravenous Infusion (IV) over 60 minutes on Days 1 and 15 (28-day cycle).
Arm/Group | Phase II Schedule C. LDAC | Phase I Schedule A. Volasertib 150 mg+LDAC | Phase I Schedule A. Volasertib 200 mg+LDAC | Phase I Schedule A. Volasertib 250 mg+LDAC | Phase I Schedule A. Volasertib 300 mg+LDAC | Phase I Schedule A. Volasertib 350 mg+LDAC | Phase II Schedule A. Volasertib 350 mg+LDAC | Phase I Schedule A. Volasertib 400 mg+LDAC | Phase I Schedule B. Volasertib 150 mg | Phase I Schedule B. Volasertib 200 mg | Phase I Schedule B. Volasertib 350 mg | Phase I Schedule B. Volasertib 400 mg | Phase I Schedule B. Volasertib 450 mg | Phase I Schedule B. Volasertib 500 mg | Phase I Schedule B. Volasertib 550 mg
All-Cause Mortality (participants affected / at risk) | 45/45 | 4/4 | 3/3 | 4/5 | 9/9 | 8/8 | 38/42 | 3/3 | 11/11 | 2/2 | 3/5 | 6/6 | 21/23 | 5/5 | 4/4
Serious Adverse Events (participants affected / at risk) | 29/45 | 2/4 | 3/3 | 3/5 | 7/9 | 6/8 | 34/42 | 3/3 | 7/11 | 1/2 | 3/5 | 3/6 | 16/23 | 3/5 | 3/4
Other Adverse Events (participants affected / at risk) | 43/45 | 4/4 | 3/3 | 5/5 | 9/9 | 8/8 | 41/42 | 3/3 | 11/11 | 2/2 | 5/5 | 6/6 | 23/23 | 5/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase II Schedule C. LDAC (N=45) | Phase I Schedule A. Volasertib 150 mg+LDAC (N=4) | Phase I Schedule A. Volasertib 200 mg+LDAC (N=3) | Phase I Schedule A. Volasertib 250 mg+LDAC (N=5) | Phase I Schedule A. Volasertib 300 mg+LDAC (N=9) | Phase I Schedule A. Volasertib 350 mg+LDAC (N=8) | Phase II Schedule A. Volasertib 350 mg+LDAC (N=42) | Phase I Schedule A. Volasertib 400 mg+LDAC (N=3) | Phase I Schedule B. Volasertib 150 mg (N=11) | Phase I Schedule B. Volasertib 200 mg (N=2) | Phase I Schedule B. Volasertib 350 mg (N=5) | Phase I Schedule B. Volasertib 400 mg (N=6) | Phase I Schedule B. Volasertib 450 mg (N=23) | Phase I Schedule B. Volasertib 500 mg (N=5) | Phase I Schedule B. Volasertib 550 mg (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 2 | 2 | 2 | 2 | 3 | 23 | 2 | 0 | 0 | 0 | 2 | 9 | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Long QT syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 5 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 2
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 8 | 0 | 0 | 1 | 0 | 0 | 5 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess neck (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspergillus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0 | 8 | 0 | 3 | 0 | 0 | 0 | 4 | 2 | 1
Pneumonia fungal (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary mycosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stenotrophomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute psychosis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheterisation venous (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase II Schedule C. LDAC (N=45) | Phase I Schedule A. Volasertib 150 mg+LDAC (N=4) | Phase I Schedule A. Volasertib 200 mg+LDAC (N=3) | Phase I Schedule A. Volasertib 250 mg+LDAC (N=5) | Phase I Schedule A. Volasertib 300 mg+LDAC (N=9) | Phase I Schedule A. Volasertib 350 mg+LDAC (N=8) | Phase II Schedule A. Volasertib 350 mg+LDAC (N=42) | Phase I Schedule A. Volasertib 400 mg+LDAC (N=3) | Phase I Schedule B. Volasertib 150 mg (N=11) | Phase I Schedule B. Volasertib 200 mg (N=2) | Phase I Schedule B. Volasertib 350 mg (N=5) | Phase I Schedule B. Volasertib 400 mg (N=6) | Phase I Schedule B. Volasertib 450 mg (N=23) | Phase I Schedule B. Volasertib 500 mg (N=5) | Phase I Schedule B. Volasertib 550 mg (N=4)
Anaemia (Blood and lymphatic system disorders) | 12 | 1 | 2 | 4 | 6 | 3 | 14 | 1 | 4 | 2 | 5 | 4 | 11 | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 0 | 0 | 0 | 1 | 0 | 8 | 0 | 1 | 0 | 1 | 0 | 4 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 1 | 1 | 2 | 5 | 1 | 1 | 1 | 2 | 1 | 1 | 2 | 7 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 5 | 0 | 2 | 1 | 1 | 0 | 11 | 0 | 2 | 1 | 1 | 3 | 12 | 1 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 0 | 2 | 4 | 5 | 3 | 9 | 1 | 5 | 1 | 3 | 2 | 12 | 1 | 2
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac valve disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiomegaly (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Heart valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Adrenal disorder (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Macular degeneration (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 0 | 0 | 2 | 2 | 1 | 4 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1 | 1 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 12 | 0 | 3 | 2 | 2 | 3 | 18 | 0 | 3 | 1 | 0 | 1 | 6 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 11 | 2 | 2 | 2 | 4 | 1 | 13 | 0 | 1 | 0 | 2 | 3 | 6 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Gingival discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 16 | 2 | 0 | 2 | 4 | 4 | 19 | 2 | 2 | 0 | 0 | 1 | 7 | 2 | 2
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestine ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 5 | 3 | 0
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 2 | 1 | 1 | 4 | 0 | 16 | 1 | 1 | 1 | 0 | 0 | 6 | 1 | 1
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 11 | 0 | 0 | 1 | 1 | 0 | 10 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Calcinosis (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site erythema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 3 | 0 | 1 | 0 | 2 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 1 | 0 | 2 | 1 | 3 | 2 | 2 | 1 | 0 | 1 | 0 | 1 | 2 | 0
Fatigue (General disorders) | 11 | 1 | 1 | 5 | 5 | 4 | 11 | 1 | 3 | 2 | 1 | 0 | 4 | 2 | 2
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Feeling of body temperature change (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 1 | 2 | 1 | 3 | 5 | 1 | 1 | 0 | 1 | 2 | 13 | 1 | 0
Granuloma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Induration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 2 | 0 | 0 | 1 | 2 | 3 | 10 | 0 | 1 | 0 | 1 | 2 | 2 | 0 | 0
Oedema (General disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 1
Oedema mucosal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 9 | 0 | 2 | 1 | 5 | 2 | 12 | 1 | 2 | 1 | 1 | 1 | 9 | 0 | 0
Pain (General disorders) | 3 | 1 | 0 | 0 | 1 | 3 | 5 | 1 | 3 | 0 | 1 | 1 | 3 | 0 | 0
Puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 8 | 0 | 1 | 1 | 4 | 1 | 13 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Thirst decreased (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic congestion (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic lesion (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fusobacterium infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Micrococcus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nail bed infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 1 | 2 | 4 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Drug administration error (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 4 | 1 | 4 | 1 | 0 | 0 | 0 | 1 | 4 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 1
Activated partial thromboplastin time shortened (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 4 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 5 | 1 | 0
Blast cell count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood albumin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 0
Blood chloride increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 3 | 1 | 0 | 1 | 3 | 1 | 2 | 0 | 2 | 1 | 2 | 2 | 6 | 0 | 2
Blood fibrinogen increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Blood iron decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood iron increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 3 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 3 | 1 | 1 | 2 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 1
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 5 | 2 | 1 | 2 | 4 | 4 | 2 | 1 | 4 | 2 | 1 | 3 | 7 | 1 | 3
Candida test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 1
Electrocardiogram change (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterococcus test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 4 | 0 | 1 | 0 | 3 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatic specific antigen increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0
Prothrombin time prolonged (Investigations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Serum ferritin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombin time shortened (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
White blood cells urine (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 2 | 2 | 4 | 5 | 2 | 6 | 1 | 3 | 0 | 1 | 2 | 10 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 4 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 3 | 2 | 1 | 2 | 0 | 2 | 2 | 2 | 1 | 6 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 4 | 4 | 6 | 8 | 3 | 2 | 0 | 0 | 0 | 10 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 4 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Iron overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Uraemic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 0 | 3 | 1 | 7 | 0 | 0 | 0 | 1 | 0 | 3 | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 2 | 1 | 1 | 2 | 0 | 6 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 1
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 0 | 0 | 2 | 3 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Leukaemia cutis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 1 | 4 | 2 | 2 | 3 | 1 | 1 | 0 | 0 | 0 | 4 | 0 | 1
Headache (Nervous system disorders) | 7 | 1 | 0 | 0 | 0 | 1 | 4 | 1 | 1 | 0 | 2 | 1 | 5 | 2 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Orthostatic intolerance (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 1 | 1 | 1 | 5 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Communication disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bladder pain (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 2 | 2 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Micturition disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal atrophy (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urethral haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urethral pain (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast enlargement (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital swelling (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematospermia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nipple disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Penile oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal erythema (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 1 | 2 | 4 | 2 | 10 | 0 | 2 | 0 | 0 | 1 | 6 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 1 | 0 | 4 | 2 | 10 | 0 | 1 | 0 | 0 | 2 | 4 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 3 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 0 | 0 | 1 | 3 | 2 | 16 | 0 | 2 | 1 | 2 | 2 | 5 | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 5 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 4 | 1 | 3 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 1 | 0 | 0 | 1 | 3 | 3 | 0 | 2
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 1 | 0 | 0 | 4 | 1 | 1 | 0 | 1 | 3 | 3 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parapsoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 2 | 2 | 2 | 10 | 2 | 4 | 0 | 1 | 4 | 3 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 2 | 1 | 1 | 3 | 4 | 0 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fasting (Social circumstances) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Central venous catheterisation (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angiopathy (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 1 | 0 | 2 | 1 | 3 | 2 | 0 | 2 | 1 | 0 | 3 | 3 | 2 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 4 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 5 | 1 | 2
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 1 | 0 | 1 | 1 | 7 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infarction (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyphaema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palatal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital burning sensation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT00804856/Prot_000.pdf
  • Statistical Analysis Plan (2012-01-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT00804856/SAP_001.pdf